CLINICAL TRIAL: NCT02365012
Title: Treatment of Orthostatic Intolerance in Patients With Parkinson's Disease Using Midodrine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Stephanie Pawlowski Wood, Research Administrator, Corporal Michael J. Crescenz VA Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 01482
Record Dates: First submitted 2015-02-10; First posted 2015-02-18 (Estimated); Last update posted 2015-08-26 (Estimated); Status verified 2015-08

CONDITIONS: Orthostatic Intolerance; Parkinson's Disease
MeSH Terms: conditions — Orthostatic Intolerance; Parkinson Disease | interventions — Midodrine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo given three times a day for 2 weeks
- Midodrine (Active Comparator): Midodrine 2.5 mg given three times a day for one week followed by 5 mg given three times a day for one week
  Interventions: Drug: Midodrine

INTERVENTIONS:
Drug: Midodrine — Crossover intervention comparing midodrine to placebo for subjects with orthostatic intolerance
  Arms: Midodrine

SUMMARY:
This study will evaluate whether treatment with the α1-agonist, midodrine, reduces subjective orthostatic lightheadedness as measured by the Non-Motor Symptoms Scale for Parkinson's Disease (NMSS) questionnaire, in patients with (positive control group, OH) or without documented orthostatic hypotension(orthostatic intolerance, OI). It will also demonstrate the effect of treatment with an α1-agonist, midodrine, on beat-to-beat blood pressure and heart rate response during Valsalva maneuver (measured by Continuous Non-invasive Arterial Pressure, CNAP) in patients with OI or OH and evaluate the relationship to symptom improvement.

DETAILED DESCRIPTION:
This will be a cross-over study where participants with OI will be randomized to initially receive midodrine or placebo then crossed over to the opposite treatment after three weeks (2 weeks on midodrine or placebo plus one week wash out period). The control group will consist of participants with OH and PD being treated with midodrine. Basic demographic data including will be collected from the medical record of each participant after consent. At each study visit, each participant will undergo traditional measurement of blood pressure and heart rate as well as measurement of beat-to-beat blood pressure and heart rate using CNAP™ during valsalva maneuver and in response to standing for 5 minutes after sitting. Symptoms of orthostatic intolerance will be measured during the study visit using Domain 1 of the Non-Motor Symptoms Scale for Parkinson's Disease (NMSS). At the initial study visit, participants will also be administered first dose of midodrine or placebo. Supine sitting, and standing systolic and diastolic blood pressure and pulse rates will be measured immediately before and 1 hour after the administration of drug or placebo. This blood pressure monitoring process will take place at each of the four study visits.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of idiopathic Parkinson's Disease
2. Those patients with measured orthostatic hypotension will be included in the positive control group
3. Those patients without measurable orthostatic hypotension who have symptoms of lightheadedness on standing will be included in the study group

Exclusion Criteria:

1. Diagnosis of degenerative parkinsonian syndromes other than idiopathic Parkinson's Disease
2. Inability to stand independently and remain standing for 5 minutes
3. Cognitive impairment that is significant enough to affect the ability of the patient to provide informed consent or to reliably report orthostatic symptoms
4. Patients with a pacemaker will also be excluded because the study is measuring heart rate responses which could potentially be altered by a pacemaker
5. Because this study will be using a drug that can affect blood pressure, those patients with a standing BP of > 139/90 and heart rate <60 will be excluded
6. Because this study will be using a drug that can affect supine hypertension, those patients with a supine BP of >139/90 and heart rate <60 will be excluded
7. Current treatment with other drugs for orthostatic hypotension such as fludrocortisone
8. Patients on phenylephrine, pseudoephedrine, ephedrine, phenylpropanolamine, dihydroergotamine
9. Patients with acute or chronic renal failure (GFR <60)
10. Patients with a history of pheochromocytoma, urinary retention, severe cardiac disease, history of congestive heart failure, diabetes, narrow-angle glaucoma, arrhythmias, bradycardia, severe hyperthyroidism, severe difficult urination (due to urinary retention or enlarged prostate)
11. Pregnant or breast-feeding women.
12. Women of childbearing potential with no effective contraceptive method of birth control and/or who are unwilling or unable to be tested for pregnancy.
13. Women of childbearing potential must have a confirmed negative pregnancy test at screening and randomization visits. They must use an effective contraceptive method throughout the study, and agree to repeat urine pregnancy test at designated visits. The applied methods of contraception have to meet the criteria for a highly effective method of birth control (condoms, FDA approved oral contraceptives, patches, injections, rings, IUD).
14. Patients with known drug allergy or hypersensitive to midodrine.

Ages: 22 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2014-04; Primary Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
NMSS Domain I (improvement in symptoms of lightheadedness when standing) | 7 weeks
  improvement in symptoms of lightheadedness when standing

SECONDARY OUTCOMES:
Valsalva response (Beat-to-beat blood pressure and heart rate variation during Valsalva maneuver) | 7 weeks
  Beat-to-beat blood pressure and heart rate variation during Valsalva maneuver

CONTACTS AND LOCATIONS:
Overall Officials: James Morley, DOMD/Ph.D., Principal Investigator — PVAMC
Locations (1):
- PVAMC, Philadelphia, Pennsylvania, United States